CLINICAL TRIAL: NCT04882683
Title: Clinical Study of Cord Blood Mononuclear Cells on Treatment of Hormone-resistant or Hormone-dependent Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB-MNCs-UC-2021
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; umbilical cord blood mononuclear cells; safety and efficacy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Prednisone; Azathioprine; Adalimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Prednisone+Azathioprine/Adalimumab
  Interventions: Drug: Prednisone; Drug: Azathioprine; Drug: Adalimumab
- UCB-MNCs group (Experimental): Prednisone+Azathioprine/Adalimumab+UCB-MNCs
  Interventions: Drug: Prednisone; Drug: Azathioprine; Drug: Adalimumab; Biological: umbilical cord blood mononuclear cells

INTERVENTIONS:
Drug: Prednisone — 0.75 mg per kilogram per day for three months
  Other Names: Deltacortone; Meticorten
Drug: Azathioprine — 1 mg per kilogram per day for three months
  Other Names: Imurek; Imurel
Drug: Adalimumab — 40mg every two weeks for three months
  Other Names: Humira
Biological: umbilical cord blood mononuclear cells — Peripheral intravenous infusion method, infusion of umbilical cord blood mononuclear cell suspension 50ml (cell number 2×10^8).
  Arms: UCB-MNCs group

SUMMARY:
This study conducted a systematic clinical observation of the clinical efficacy of UCB-MNCs in the treatment of hormone-resistant or hormone-dependent ulcerative colitis, in order to observe its clinical safety and efficacy.

DETAILED DESCRIPTION:
This study adopts a randomized and controlled clinical research design. Patients are randomly divided into conventional treatment control group and UCB-MNCs treatment test group. The control group is given conventional treatment: prednisone combined azathioprine or adalimumab; the test group is given conventional treatment combined UCB-MNCs treatment, follow-up observations were carried out, in order to observe the clinical efficacy and safety of UCB-MNCs in the treatment of hormone resistance or hormone-dependent ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Western medicine diagnosis is consistent with patients with refractory ulcerative colitis.
* 2. 18 Years to 65 Years，male or female.
* 3. Those who voluntarily participate in this clinical study and have signed an informed consent.

Exclusion Criteria:

* 1. Patients with non-refractory UC.
* 2. Those who are pregnant or breastfeeding, or have a childbirth plan in the near future.
* 3. People with severe allergies or allergies to known ingredients in basic treatments.
* 4. Patients with severe primary diseases such as severe cardiovascular and cerebrovascular diseases, liver and kidney, and hematopoietic system.
* 5. There are serious complications, such as local stenosis, intestinal obstruction, intestinal perforation, multiple intestinal polyps, toxic megacolon, rectal cancer, etc..
* 6. Patients with mental disorders and intellectual disabilities.
* 7. Patients who have participated in clinical studies of other drugs in the past 3 months.
* 8. Those who are seriously ill and need emergency treatment.
* 9. Patients who are still undergoing other treatment options for ulcerative colitis.
* 10. Researchers believe that it is not suitable for entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy rate | Change from Baseline Clinical efficacy rate at 8th and 16th week, and the first week after the end of treatment.
  According to the method of modified Mayo score calculation, it is defined as a decrease of ≥30% of the score or a decrease of ≥3 points relative to the baseline value, and a decrease of ≥1 point or a score of 0 or 1 in the sub-item score of blood in the stool, and this type of patient is judged Effective for treatment. Clinical effective rate = (effective number of people / total number of people in this group ) × 100%.
Clinical response rate | Change from Baseline Clinical response rate at 8th and 16th week, and the first week after the end of treatment.
  According to the method of modified Mayo score calculation, it is defined as a score ≤ 2 points and no single sub-item score> 1 point. Clinical remission rate =(number of remissions / total number of people in this group) × 100%.

SECONDARY OUTCOMES:
Clinical symptom score | Change from Baseline clinical symptom score at the first week after the end of treatment.
  According to the scoring criteria for individual symptoms (diarrhea, mucus pus and blood in the stool, abdominal pain, tenesmus), the severity of symptoms is divided into 0, 2, 4, and 6 points. The higher the score, the more severe the symptoms.
Endoscopic response rate | Change from Baseline endoscopic response rate at the first week after the end of treatment.
  According to the method of modified Mayo score, endoscopy found that the score decreased by at least 1 point from baseline. Endoscopic response rate = (number of endoscopic responders/total number of people in the group) × 100%.
Mucosal healing rate | Change from Baseline mucosal healing rate at the first week after the end of treatment.
  According to the method of modified Mayo score, the absolute score of the endoscopy discovery score is 0 or 1 point. Mucosal healing rate = (mucosal healing number / total number of people in this group) × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Shandong, Shandong, China

IPD SHARING:
Plan to Share IPD: No